CLINICAL TRIAL: NCT00953277
Title: A Pilot Study to Assess the Technical Feasibility of Robotic Assisted Laparoscopic Interpositioning of the AVANCETM Nerve Graft for Reconstruction of the Neurovascular Bundle, With a Twenty-four Month Follow-up Term to Assess Efficacy
Brief Title: Study of Nerve Reconstruction Using AVANCE in Subjects Who Undergo Robotic Assisted Prostatectomy for Treatment of Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANG-CP-003
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Nerve Injury; Prostate Cancer; Radical Prostatectomy; Nerve Reconstruction; Cavernous Nerve Injury
Keywords: Nerve Repair; Erectile Function; Prostate Cancer; Robot Assisted Laparoscopic Prostatectomy; Continence
MeSH Terms: conditions — Peripheral Nerve Injuries; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avance Nerve Graft (Experimental): Processed Human Nerve Tissue Scaffold
  Interventions: Other: Processed Human Nerve Tissue Scaffold

INTERVENTIONS:
Other: Processed Human Nerve Tissue Scaffold — Implantation of appropriate length of processed human nerve scaffold at the time of surgery.

SUMMARY:
The purpose of this study is to determine if it is technically feasable to repair nerves that are injured as part of a planned surgical removal of the prostate and the surrounding tissue in subjects with prostate cancer. The study will also examine the long term outcomes on erectile function, continence and overall quality of life in the enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, but ≤70 years of age;
* IIEF EF Domain*1 score ≥ 22;
* be able to effectively communicate with study personnel;
* be considered by the physician to be available for subsequent visits;
* be willing to comply with all aspects of the treatment and evaluation schedule over a 24 month duration;
* sign and date an IRB-approved written informed consent prior to initiation of any study procedures, including screening procedures; and
* require radical prostatectomy.

Exclusion Criteria:

* prior surgery in the last 6 months which could affect sexual function;
* history of Peyronie's disease;
* significant neurological disorder (i.e. multiple sclerosis, peripheral neuropathy);
* treatment for major psychiatric disorders;
* history of penile implant or prosthesis;
* history of diabetic neuropathy;
* life expectancy of less than two years;
* concurrently involved in another investigational study;
* uncontrolled hypertension with systolic BP >200mmHg or diastolic BP >115mmHg is present at screening;
* currently receiving or planned treatment with chemotherapy or radiation therapy;
* diagnosis of bony metastasis;
* known allergy or severe intolerance to PDE-5 inhibitors; or
* cardiac pacing equipment or other electro-mechanical devices which preclude the use of CaverMap™ neurostimulator.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Surgeon Assessment of Technical Feasibility | At time of surgery

SECONDARY OUTCOMES:
Erectile Recovery Rates | Month 1, 3, 6, 9, 12, 18 and 24
Continence Rates | Month 1, 3, 6, 9, 12, 18 and 24
Quality of Life Questionnaire | Month 1, 3, 6, 9, 12, 18 and 24
Adverse Events | Month 1, 3, 6, 9, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Smith, MD, Principal Investigator — Vanderbilt Univerisity
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States